CLINICAL TRIAL: NCT00236379
Title: A Six-month, Double-blind, Randomized, International, Multicenter Trial to Evaluate the Glucoregulatory Effects of Risperidone and Olanzapine in Subjects With Schizophrenia or Schizoaffective Disorder
Brief Title: A Study of the Effects of Risperidone and Olanzapine on Blood Glucose (Sugar) in Patients With Schizophrenia or Schizoaffective Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen, LP (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002758
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-03

CONDITIONS: Schizophrenia; Diabetes Mellitus
Keywords: schizophrenia; blood glucose; glucose metabolism; diabetes mellitus; risperidone; olanzapine
MeSH Terms: conditions — Schizophrenia; Diabetes Mellitus | interventions — Olanzapine; Risperidone

ARMS (2):
- 001 (Experimental): Risperidone Target oral dose of 6 milligrams per day for for 6 months
  Interventions: Drug: Risperidone
- 002 (Experimental): Olanzapine Target oral dose of 20 milligrams per day for 6 months
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine — Target oral dose of 20 milligrams per day for 6 months
  Arms: 002
Drug: Risperidone — Target oral dose of 6 milligrams per day for for 6 months
  Arms: 001

SUMMARY:
The purpose of this study is to assess and compare how risperidone and olanzapine, two antipsychotic medications, affect the regulation of glucose (sugar) in the body.

DETAILED DESCRIPTION:
The newer antipsychotic medications risperidone and olanzapine effectively treat schizophrenia and related disorders, and they may cause fewer side effects than the older antipsychotic drugs do. However, some of the newer antipsychotic medications could have a negative effect on the regulation of blood glucose (sugar) in the body. This negative effect could make the patient gain weight and even develop diabetes mellitus. This randomized, double-blind study will assess and compare how risperidone and olanzapine affect the regulation of glucose in the body in patients with schizophrenia and schizoaffective disorder. Patients will be randomly assigned to receive risperidone (target oral dose of 6 milligrams per day) or olanzapine (target oral dose of 20 milligrams per day) for 6 months. Repeat laboratory measurements will be performed and questions will be asked of the patients to evaluate the safety and effectiveness of the drugs. The primary laboratory test used to assess the patient's regulation of blood glucose will be the Disposition Index derived from the Frequently Sampled Intravenous Glucose Tolerance Test. Risperidone 2 milligram oven-encapsulated tablets taken orally once a day for 6 months; olanzapine 5 milligram tablets taken orally once a day for 6 months

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or related disorder
* stable with respect to disease symptoms and other medical conditions
* would benefit from this type of antipsychotic drug
* if female, using birth control.

Exclusion Criteria:

* Patients who are delirious, bipolar, severely mentally retarded, or suicidal
* psychiatric diagnosis of disease unrelated to schizophrenia
* presence of stroke, brain tumor, Parkinson's Disease, or diseases that affect blood glucose control
* history of diabetes
* long or recent history of taking risperidone, olanzapine, quetiapine, clozapine, or investigational drugs
* recent history of unstable thyroid function
* if female, not using birth control
* abusing drugs or alcohol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Change in the Disposition Index derived from the Frequently Sampled Intravenous Glucose Tolerance Test (which shows how the body regulates glucose) | Up to 6 months

SECONDARY OUTCOMES:
Changes in measurements of metabolism and glucose regulation; changes in results of tests and questionnaires evaluating the effectiveness and safety (including laboratory tests and anthropomatic measurements) of medications used to treat schizophrenia | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Janssen, LP Clinical Trial, Study Director — Janssen, LP

REFERENCES:
- See also: A Six-Month, Double Blind, Randomized, International, Multicenter Trial to Evaluate the Glucoregulatory Effects of Risperidone and Olanzapine in Subjects with Schizophrenia or Schizoaffective disorder. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=345&filename=CR002758_CSR.pdf